CLINICAL TRIAL: NCT06579638
Title: Patterns and Outcomes of Peripheral Vascular Complications Following Self-injection of Addictive Drugs.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Marghny Hassan, Resident, Assiut University
Other Study IDs: IVDA Complications
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: IVDA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intravascular drug abuse is a common health problem with increasing prevalence throughout the world. The estimated number of IV drug abusers around the world is15.6 millions.

DETAILED DESCRIPTION:
Intravascular drug abuse is a common health problem with increasing prevalence throughout the world. The estimated number of IV drug abusers around the world is15.6 millions.The prevalence of injected drug use is estimated between 0.09% and 1.3% depending on geographic location. There are various complications of IV drug abuse that are related to the toxicity of the substance, mode of consumption, and drug taking mode. These complications include skin and soft tissue infection (cellulitis, abscess, necrotizing fasciitis) (28%),infected(ranges from .03% to 1%)or non-infected pseudoaneurysm ,arterial ischemia( thrombosis , distal embolization), and venous thrombosis(29%).

The wide spectrum of complications due to IVDA mandates a wide range of treatment for each type starting from simple medical treatment such as antibiotics or anticoagulation to the most extensive surgical treatment options in cases such as PA that may require ligation of the arterial supply without revascularization. This may lead to gravid complications such as limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* Current IV drug abuser
* (Age from 18 to 80 )
* Presented with peripheral vascular complications (pseudoaneurysm, limb ischemia, venous thrombosis, skin infection.)

Exclusion Criteria:

* Drug intake other than IV
* ( less than 18 or more than 80 )
* Presented with overdose
* Malignancy or serious illness
* Causes of vascular complications other than IV drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients developing peripheral vascular complications due to IVDA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Patterns and outcomes of IVDA | 1 year
  To describe the patterns, methods of treatment and outcomes of self-injection of addictive drugs such as amputation rate and patency rate.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa S Khalil, Professor, Study Chair — Assiut University; Ashraf G Taha, Assist. prof, Study Director — Assiut University; Mohamed S Abdelkareem, Lecturer, Study Director — Assiut University; Islam M Hassan, Resident, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsao JW, Marder SR, Goldstone J, Bloom AI. Presentation, diagnosis, and management of arterial mycotic pseudoaneurysms in injection drug users. Ann Vasc Surg. 2002 Sep;16(5):652-62. doi: 10.1007/s10016-001-0124-6. Epub 2002 Sep 4. PMID 12203000
- [Result] Senbanjo R, Strang J. Evaluation of Femoral Ultrasonography as a Tool for Promoting Cessation of Groin-Injecting Behaviour. Eur Addict Res. 2015;21(4):204-10. doi: 10.1159/000375260. Epub 2015 Apr 21. PMID 25896872
- [Result] Degenhardt L, Peacock A, Colledge S, Leung J, Grebely J, Vickerman P, Stone J, Cunningham EB, Trickey A, Dumchev K, Lynskey M, Griffiths P, Mattick RP, Hickman M, Larney S. Global prevalence of injecting drug use and sociodemographic characteristics and prevalence of HIV, HBV, and HCV in people who inject drugs: a multistage systematic review. Lancet Glob Health. 2017 Dec;5(12):e1192-e1207. doi: 10.1016/S2214-109X(17)30375-3. Epub 2017 Oct 23. PMID 29074409